CLINICAL TRIAL: NCT05793632
Title: Role of Quetiapine in the Prevention of ICU Delirium in Elderly Patients at a High Risk
Brief Title: Quetiapine in Prevention of Delirium
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Quetiapine
Record Dates: First submitted 2023-02-28; First posted 2023-03-31 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-03

CONDITIONS: Delirium
MeSH Terms: conditions — Delirium | interventions — Quetiapine Fumarate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Quetiapine (Experimental): The patients with multiple risks for delirium will receive 25 mg/day PO
  Interventions: Drug: Quetiapine
- Non pharmacological preventive bundle (No Intervention): The patients will only be monitored with application of delirium preventive bundle without pharmacological agent

INTERVENTIONS:
Drug: Quetiapine — The patients will be randomly divided into two equal groups group Q and group C. Randomization will be done by computer-generated number lists and using opaque sealed envelopes.
  Arms: Quetiapine

SUMMARY:
The aim is to study the effectiveness of Quetiapine in preventing delirium in the elderly patients with multiple risks for delirium.

ELIGIBILITY:
Inclusion Criteria:

* Patients with anemia
* Sedated patients
* Hypotensive patients
* Immobilized patients
* Patients with visual or auditory impairment

Exclusion Criteria:

* Patients or guardians refuse to participate
* Patients diagnosed with delirium
* Contraindication for delirium

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-15 (Actual)

PRIMARY OUTCOMES:
Quetiapine in preventing delirium | 2 months
  The presence of delirium will be monitored among the patients in the two groups using ICU-Confusion Assessment Method 7 score for delirium where a score of (0-2 = no delirium, 3-5 = mild to moderate delirium and a score >5 = severe delirium)

CONTACTS AND LOCATIONS:
Overall Officials: Walid Kamel, Principal Investigator — Faculty of medicine, Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Egypt